CLINICAL TRIAL: NCT03536195
Title: Impact of Renal Replacement Therapy on Coagulation Profile in Patients with Acute Renal Failure
Brief Title: Impact of Renal Replacement Therapy on Coagulation Profile of Patients with Acute Renal Failure
Acronym: HEMOSTIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: HEMOSTIR (29BRC17.0132)
Record Dates: First submitted 2018-04-25; First posted 2018-05-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Acute Renal Failure; Hemorrhage; Coagulation Disorder
Keywords: renal replacement therapy; acute renal failure; coagulation; bleeding
MeSH Terms: conditions — Acute Kidney Injury; Hemorrhage; Hemostatic Disorders; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Renal failure and high plasmatic level of urea have been associated with an increased risk of hemorrhage in surgical patients. There is only sparse data on the impact of renal replacement therapy on homeostatic parameters. The aim of this study is to describe potential changes in homeostatic parameters before and after renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients
* acute renal failure
* renal replacement therapy
* plasmatic urea > 20

Exclusion Criteria:

* chronic renal failure
* platelet count less than 80 Giga
* V factor less than 70%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with acute renal failure where the decision of renal replacement therapy has been made.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-08-18 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
visco elastometry | Change in ROTEM parameters from baseline to after renal replacement therapy
  ROTEM (Rotational Thromboelastometry)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No